CLINICAL TRIAL: NCT00996970
Title: Immunogenicity of Novel H1N1 Vaccination Among HIV-Infected Compared to HIV-Uninfected Persons
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Infectious Diseases Clinical Research Program (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IDCRP-053
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Influenza; HIV Infections
Keywords: HIV; H1N1; Influenza; Vaccination; Seroresponse; Immunogenicity; Vaccine
MeSH Terms: conditions — Influenza, Human; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for immunologic studies including antibody titers and cellular responses. Viral isolates will be obtained and characterized among ILI cases during study participation. Blood for CD4/HIV RNA levels will also be obtained among HIV patients to determine the impact of the vaccine on these counts.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to determine the effectiveness of the novel H1Nl influenza (inactivated/killed formulation) vaccine among both HIV-infected and HIV-uninfected persons. The administration of the H1Nl vaccination is not part of the study's procedures, but is being given as part of routine care.

DETAILED DESCRIPTION:
The investigators study is being conducted to evaluate and compare the seroresponses of the novel H1N1 vaccination among HIV positive and negative persons receiving the novel H1N1 vaccination as part of routine clinical care, with secondary objectives examining the impact of prior seasonal vaccinations on subsequent seroresponse to the novel H1N1 vaccination, determining potential reactions (local or systemic) to this new vaccine among patients, and assessing for potential immunologic/virologic changes (in CD4/HIV RNA levels) after H1N1 vaccination among HIV patients. Finally, the investigators will collect data on influenza-like illnesses (ILI) and H1N1 events during the study follow-up period and influenza isolates causing ILI events will be genetically characterized.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Receiving the novel H1N1 vaccine (killed formulation) as part of routine clinical care
* A military beneficiary who expects to remain in the local area for the next 6 months

Exclusion Criteria:

* Healthcare worker who is involved in direct patient care
* Acute febrile illnesses within 30 days prior to H1N1 vaccination (e.g., pneumonia, influenza, ILI)
* Diabetes type 1 or type 2
* Systemic steroid or immunosuppressive medication use within 4 weeks of vaccination
* Active diagnoses of a cancer (non-melanoma skin cancer allowed).
* History of organ transplant
* Chronic active hepatitis B or C
* Active illicit drug use or alcohol abuse
* Blood transfusion within the last year
* Allergy to eggs
* Previous significant adverse reaction (e.g., anaphylaxis) to the seasonal influenza vaccination
* History of serious reactions to any prior vaccination (e.g., Guillain Barre Syndrome (GBS)).
* Received another vaccination in the last 4 weeks (receipt of seasonal influenza vaccination is allowed)
* Among females of childbearing potential, pregnant or within 6 weeks of being postpartum
* History of ILI which was confirmed as an H1N1 infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Males and females of all races and all military beneficiaries including active duty enlisted and officers (from all branches of service), retirees, and their dependents presenting for H1N1 vaccination as part of routine clinical care will be eligible for participation. Both HIV-positive and negative persons can participate. Since most of our HIV patients are 18-50 years of age, and seroresponse varies by age, we will enroll persons between the ages of 18-50 years.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
To compare the immunogenicity via anti-hemagglutinin responses following H1N1 vaccination between HIV positive and negative persons. | interim = 2 months; 6 month f/u = 8 months

SECONDARY OUTCOMES:
To compare the immunogenicity via HAI titer levels, microneutralization seroresponses and titer levels, and cellular responses following H1N1 vaccination between HIV positive and negative persons. | 1 year
Among those undergoing vaccination with the seasonal influenza vaccine during the current influenza season, to compare the presence of a positive seroresponse between HIV positive and negative persons | 1 year
To evaluate the effect of pre-existing anti-influenza immunity and recent history of seasonal influenza vaccination on seroresponses to the H1N1 influenza vaccine among both HIV positive and negative persons. | 1 year
To compare the durability of the H1N1 immunologic responses at 6 months post-vaccination between HIV-infected and uninfected persons. | 1 year
To evaluate the number of ILIs and documented influenza cases among HIV-infected and uninfected persons after initial vaccination, and to genetically characterize the influenza strains causing ILI events in our study cohort. | 1 year
To evaluate the impact of CD4 counts/percentages, HIV RNA levels, and HAART use on the immunologic responses to H1N1 vaccination in HIV positive subjects. | 1 year
To evaluate the impact of the H1N1 vaccine on CD4 counts/percentages and HIV RNA levels in HIV positive subjects. | 2 months
To evaluate potential adverse reactions of the H1N1 vaccine in HIV positive versus negative subjects. | 2 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Naval Medical Center Portsmouth, Portsmouth, Virginia

REFERENCES:
- [Derived] Crum-Cianflone NF, Eberly LE, Duplessis C, Maguire J, Ganesan A, Faix D, Defang G, Bai Y, Iverson E, Lalani T, Whitman T, Blair PJ, Brandt C, Macalino G, Burgess T. Immunogenicity of a monovalent 2009 influenza A (H1N1) vaccine in an immunocompromised population: a prospective study comparing HIV-infected adults with HIV-uninfected adults. Clin Infect Dis. 2011 Jan 1;52(1):138-46. doi: 10.1093/cid/ciq019. Epub 2010 Dec 7. PMID 21148532